CLINICAL TRIAL: NCT03213886
Title: A Prospective Randomized Trial Comparing the Effects of 2 Vitamin D Supplementation Regimens in Elderly People After Hip Fracture Surgery
Brief Title: The Effect of Supplementation of Vitamin D Deficiency in Older People With Acute Hip Fracture:
Acronym: VITAMINA_D
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Leonor Cuadra Llopart (Other)
Collaborators: Fundacio Salut i Envelliment UAB (Other)
Responsible Party: Sponsor-Investigator, Leonor Cuadra Llopart, Medical Doctor, Consorci Sanitari de Terrassa
Organization: Consorci Sanitari de Terrassa (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VITAMINA_D; 2017-001778-40 (EudraCT Number)
Record Dates: First submitted 2017-06-27; First posted 2017-07-11 (Actual); Last update posted 2021-02-02 (Actual); Status verified 2021-01

CONDITIONS: Hip Fracture; Vitamin D Deficiency
Keywords: hip fracture; elderly; vitamin D; rehabilitation
MeSH Terms: conditions — Hip Fractures; Vitamin D Deficiency | interventions — Calcifediol; Vitamin D

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Calcifediol (Vitamin D) loading-dose (Experimental): Participants in the intervention group will receive calcifediol16.000 units (U) /day for five days
  Interventions: Drug: Calcifediol (Vitamin D)
- Calcifediol (Vitamin D) at clinical practice dose (Active Comparator): Participants in the control group will receive 16.000 U / week for five weeks
  Interventions: Drug: Calcifediol (Vitamin D)

INTERVENTIONS:
Drug: Calcifediol (Vitamin D) — After surgical treatment, participants with vitamin D deficiency (25OHD < 30 ng/mL) will be randomly allocated to an intervention group or control group.
  For the intervention group, participants will receive 16. 000 U oral Calcifediol daily for 5 days.
  For the control group, participants will receive 16.000 U oral Calcifediol weekly for 5 weeks.
  Both groups:
  1. Will follow the usual hip fracture rehabilitation pathway.
  2. 25OHD serum levels will be measured after 4 weeks. Depending on the serum 25OHD level, the patients will receive different vitamin D strategies (according to the protocol) Patients will be monitored for up to 12 months after the discharge from the hospital, with 3 clinic visits at 3, 6 and 12 months (to determine serum vitamin D levels and to evaluate functional status)

SUMMARY:
This study will be done to evaluate the effect of load dose of vitamin D compared to the dose of usual clinical practice, in improving mobility and reducing disability in older people following a hip fracture.

DETAILED DESCRIPTION:
Hip fractures and related disabilities are important public health issues for elderly people around the world. Attending the progressive aging of the population, an increase in the number of hip fractures is expected. In fact, some studies estimate that, globally, the incidence will exceed 6 million in 2050. In Spain, approximately 33,000 hip fracture occur annually, with an overall incidence of 517 cases per 100,000 elderly people. 90% occur in people over 64 years of age and the incidence increases exponentially beyond 80 years (> 64: 97/100000 inhabitants-year;> 85: 1898/100000 inhabitants-year).

Regarding the functional prognosis, those patients who survive the episode of the fracture often suffer a functional impairment. Outcomes for people who survive hip fracture are of concern, with more than one-quarter dying within a two-year period, and most of them not recovering their previous functional level. More than 10 % of survivors will be unable to return to their previous residence.

Vitamin D deficiency (serum 25 hydroxyvitamin D, 25OHD, level < 30 ng/mL) is commonly associated with hip fracture in elderly people. Without preventive treatment, however, vitamin D deficiency following hip fracture may result in proximal muscle weakness, pain, reduced dynamic balance and performance speed.

It is not clear how much Vitamin D must be taken in order to reach the optimal level. Although the benefits of supplementing patients with at least 800 to 1000 units (U)/day Vitamin D3 may be recognized, there is little information available to guide physicians regarding the appropriate management of hip fracture patients who may be severely Vitamin D deficient, specially in acute hip fracture patients.

A randomized controlled trial, including 50 older adults (aged 75 or over) who having suffered a hip fracture and with vitamin D deficiency, will be carried out. After surgical treatment, participants with vitamin D deficiency (25OHD < 30 ng/mL) will be randomly allocated to an intervention group or control group. For the intervention group, participants will receive 16.000 U Calcifediol oral daily along 5 days. For the control group will receive 16.000 U Calcifediol oral weekly along 5 weeks.

Functional status will be evaluated using Barthel Index, as well the proportion of patients reaching an optimal level of 25OHD (> 30 ng/mL) will be determined at discharge from hospital (1 month approximately), 3, 6 and 12 months of follow up.

Secondary measures include the Timed Up and Go test, gait speed test, Short Physical Performance Battery to compare the effect of the Vitamin D supplementation strategies on functional and muscle strength scales. In addition, to measure the strength and muscle mass will be used handheld dynamometer and bioimpedance analysis respectively

ELIGIBILITY:
Inclusion Criteria: Patients aged 75 years or over with fragility hip fracture (requiring surgical treatment) and vitamin D deficiency; able to provide informed consent, either directly or via the person responsible.

Definitions:

* Fragility hip fracture: understood as such those that are produced by trauma of low intensity (for example, falls from the own height in standing or smaller)
* Vitamin D deficiency: 25OHD serum levels < 30 ng / mL

Exclusion Criteria:

* Presence of severe functional dependence prior to fracture of the femur (Barthel Index < 35 points)
* Diagnosis of dementia to a moderate degree (defined on "Global Deterioration Scale" (GDS) and "Functional Assessment Staging" (FAST), GDS-FAST > 5).
* Medical conditions that contraindicate receiving vitamin D supplementation: hypercalcemia (calcemia> 10.5 mg / dL), hyperparathyroidism; chronic renal failure with glomerular filtration rate (GFR) <30 mL / min, calcium lithiasis; pathologies with risk of hypercalcemia (tuberculosis, sarcoidosis ...), as well as pathologies involving intestinal malabsorption.
* Hypersensitivity to the active substance or to any of the excipients.
* Use of drugs that interact with the use of vitamin D and with the risk of causing hypercalcemia (phenytoin, phenobarbital, primidone, digoxin).
* Reduced life expectancy (<12 months) due to the presence of advanced concomitant or end-of-life conditions.

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 50 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2019-04-20 (Actual); Study Completion 2020-07-30 (Actual)

PRIMARY OUTCOMES:
Functional gain | at 6 months of follow up
  Defined as a 15-point improvement in the Barthel Index

SECONDARY OUTCOMES:
Improvement serum Vitamin D (25OHD) levels | at baseline, 1, 3, 6 and 12 months of follow-up.
  Defined as a vitamin D levels > 30 ng/mL
Improvement of muscle strength | at 3, 6 and 12 months of follow up.
  Using handheld dynamometer to measure (kg)
Improvement of muscle mass | at 3, 6 and 12 months of follow up.
  Using bioimpedance analysis to measure (kg)

CONTACTS AND LOCATIONS:
Locations (1):
- Consorci Sanitari de Terrassa, Terrassa, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Duque G, Daly RM, Sanders K, Kiel DP. Vitamin D, bones and muscle: myth versus reality. Australas J Ageing. 2017 Mar;36 Suppl 1:8-13. doi: 10.1111/ajag.12408. PMID 28297132
- [Background] Hill TR, Aspray TJ. The role of vitamin D in maintaining bone health in older people. Ther Adv Musculoskelet Dis. 2017 Apr;9(4):89-95. doi: 10.1177/1759720X17692502. Epub 2017 Feb 14. PMID 28382112
- [Background] Dawson-Hughes B. Vitamin D and muscle function. J Steroid Biochem Mol Biol. 2017 Oct;173:313-316. doi: 10.1016/j.jsbmb.2017.03.018. Epub 2017 Mar 22. PMID 28341251
- [Background] Laiz A, Malouf J, Marin A, Longobardi V, de Caso J, Farrerons J, Casademont J. Impact of 3-Monthly Vitamin D Supplementation Plus Exercise on Survival after Surgery for Osteoporotic Hip Fracture in Adult Patients over 50 Years: A Pragmatic Randomized, Partially Blinded, Controlled Trial. J Nutr Health Aging. 2017;21(4):413-420. doi: 10.1007/s12603-016-0773-3. PMID 28346568
- [Background] Mak JC, Mason RS, Klein L, Cameron ID. An initial loading-dose vitamin D versus placebo after hip fracture surgery: randomized trial. BMC Musculoskelet Disord. 2016 Aug 11;17:336. doi: 10.1186/s12891-016-1174-9. PMID 27515154
- [Background] Sprague S, Petrisor B, Scott T, Devji T, Phillips M, Spurr H, Bhandari M, Slobogean GP. What Is the Role of Vitamin D Supplementation in Acute Fracture Patients? A Systematic Review and Meta-Analysis of the Prevalence of Hypovitaminosis D and Supplementation Efficacy. J Orthop Trauma. 2016 Feb;30(2):53-63. doi: 10.1097/BOT.0000000000000455. PMID 26429406
- [Derived] Cuadra-Llopart L, Salva Casanovas A, Cerda Mas G, Jovell-Fernandez E. Efficacy of two calcifediol supplementation regimens in older adults post-hip fracture surgery. A clinical trial. Eur Geriatr Med. 2025 Sep 15. doi: 10.1007/s41999-025-01303-y. Online ahead of print. PMID 40952661